CLINICAL TRIAL: NCT03720249
Title: Supplementation of Compound Nutrients on Plasma Homocysteine in Chinese Adults With Hyperhomocysteinemia: a Randomized Double-blind Control Trial
Brief Title: Effects of Supplementation of Compound Nutrients on Plasma Homocysteine in Chinese Adults With Hyperhomocysteinemia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Huilian Zhu (Other)
Responsible Party: Sponsor-Investigator, Huilian Zhu, professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: MN-2018-10
Record Dates: First submitted 2018-10-24; First posted 2018-10-25 (Actual); Last update posted 2019-05-14 (Actual); Status verified 2019-05

CONDITIONS: Hyperhomocysteinemia
MeSH Terms: conditions — Hyperhomocysteinemia | interventions — Betaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- supplementation of compound nutrients (Experimental): Betaine、(6S)-5-methyltetrahydrofolic acid、vitamin B6、vitamin B12 and zinc are provided as a 800mg tablet. And the tablet is orally taken once a day, four tablets at a time for 12 weeks.
  Interventions: Dietary Supplement: supplementation of compound nutrients
- placebo control (Placebo Comparator): The placebo is an excipient and the color, flavor, shape, taste and weight are same with the tablet of betaine、(6S)-5-methyltetrahydrofolic acid、vitamin B6、vitamin B12 and zinc supplement.
  Interventions: Dietary Supplement: placebo control

INTERVENTIONS:
Dietary Supplement: supplementation of compound nutrients — Betaine、 (6S)-5-methyltetrahydrofolic acid、vitamin B6、vitamin B12 and zinc per day orally for 12 weeks.
  Other Names: Betaine、 (6S)-5-methyltetrahydrofolic acid、vitamin B6、vitamin B12 and zinc supplement
  Arms: supplementation of compound nutrients
Dietary Supplement: placebo control — The placebo is an excipient and the color, flavor, shape, taste and weight are same with the tablet of supplement.
  Arms: placebo control

SUMMARY:
The purpose of this study is to determine whether supplementation of compound nutrients,including folic acid, vitamin B6, vitamin B12, betaine and zinc, will decrease the level of plasma homocysteine in Chinese adults with hyperhomocysteinemia.

ELIGIBILITY:
Inclusion Criteria:

1. People aged 18-65 years.
2. The level of plasma homocysteine is 15-100μmol/L.
3. Free from products which could decrease plasma homocysteine for at least one month.
4. Willing to participate in the study, consume the test product and perform all measurements.

Exclusion Criteria:

1. pregnant or lactating women.
2. severe diseases need to control.
3. people who unconsciousness and can not complete questionnaire.
4. long-term regular use of vitamin or mineral supplements.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-05-20 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
levels of homocysteine | 12 weeks
  At baseline, 4 weeks and 12 weeks, blood samples will be drawn and levels of homocysteine will be tested in two groups.

SECONDARY OUTCOMES:
levels of 5-methyltetrahydrofolic acid, vitamin B6, vitamin B12 and betaine | 12 weeks
  At baseline, 4 weeks and 12 weeks, blood samples will be drawn and levels of 5-methyltetrahydrofolic acid, vitamin B6, vitamin B12 and betaine will be tested in two groups.
levels of s-adenosyl-methionine and s-adenosyl-homocysteine | 12 weeks
  At baseline, 4 weeks and 12 weeks, blood samples will be drawn and levels of s-adenosyl-methionine (SAM) and s-adenosyl-homocysteine (SAH) will be tested in two groups.
anthropomorphic measurements and blood biochemical markers | 12 weeks
  Anthropomorphic measurements such as height, weight, waist circumference, hip circumference, vascular endothelial function, cardiopulmonary function, body composition and so on, and blood biochemical markers such as overnight fasting serum total cholesterol (TC), triglyceride (TG), LDL cholesterol (LDLc), HDL cholesterol (HDLc), fasting blood glucose and so on will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Huilian Zhu, professor, Study Chair — Sun Yat-sen University
Locations (1):
- SunYat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Lu XT, Wang YN, Mo QW, Huang BX, Wang YF, Huang ZH, Luo Y, Maierhaba W, He TT, Li SY, Huang RZ, Yang MT, Liu XZ, Liu ZY, Chen S, Fang AP, Zhang XG, Zhu HL. Effects of low-dose B vitamins plus betaine supplementation on lowering homocysteine concentrations among Chinese adults with hyperhomocysteinemia: a randomized, double-blind, controlled preliminary clinical trial. Eur J Nutr. 2023 Jun;62(4):1599-1610. doi: 10.1007/s00394-023-03087-y. Epub 2023 Jan 30. PMID 36717385